CLINICAL TRIAL: NCT01975688
Title: An Open-label Clinical Trial to Compare the Pharmacokinetics of up to 4 Single Oromucosal Doses of 4 Sprays of Sativex® in Patients With Treatment Induced Mild, Moderate and Severe Oral Mucositis (Grade 1 - 3 RTOG Oral Mucositis) With Their Pharmacokinetic Profile Pre-treatment (When Mucositis-free)
Brief Title: A Pharmacokinetic Study of Single Doses of Sativex in Treatment-induced Mucositis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: GW Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Organization: GWPharm (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWCP10115
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sativex: pre-treatment (Grade 0) (Experimental): The PKs of a single dose of Sativex are investigated in subjects with mucositis of Radiation Therapy Oncology Group (RTOG) Grade 0 (i.e. at baseline, pre-induction of mucositis).
  Interventions: Drug: Sativex
- Sativex: mild mucositis (Grade 1) (Experimental): The PKs of a single dose of Sativex are investigated in the same subjects when their mucositis is RTOG is Grade 1 (mild).
  Interventions: Drug: Sativex
- Sativex: moderate mucositis (Grade 2) (Experimental): The PKs of a single dose of Sativex are investigated in the same subjects when their mucositis is RTOG is Grade 2 (moderate).
  Interventions: Drug: Sativex
- Sativex: severe mucositis (Grade 3) (Experimental): The PKs of a single dose of Sativex are investigated in the same subjects when their mucositis is RTOG is Grade 3 (severe).
  Interventions: Drug: Sativex

INTERVENTIONS:
Drug: Sativex — Oromucosal spray containing THC (27 mg/mL) and CBD (25 mg/mL) in ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring.
  Each vial contains 10 mL; each 100 uL actuation delivers 2.7 mg THC and 2.5 mg CBD.
  Other Names: THC/CBD spray; Nabiximols; GW-1000-02

SUMMARY:
To investigate what the body does to single doses of Sativex (i.e. the pharmacokinetics [PKs] of four sprays containing 10.8 mg Δ9 tetrahydrocannabinol [THC] and 10 mg cannabidiol [CBD]) when mild, moderate or severe oral mucositis is induced. This will be done by looking at the effects of the body on the drug before and after oral mucositis is induced. The study participants will have Non-surgical Head and Neck Squamous Cell Carcinoma (HNSCC), and oral mucositis will be induced with radiotherapy and/or chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to give informed consent for participation in the study.
* Male or female subjects aged 18 years or above.
* Subject is diagnosed with Stage III or Stage IV HNSCC.
* Subject is due to undergo radiotherapy of the head and/or neck with or without concomitant chemotherapy with a likelihood (in the investigator's opinion) of developing mild, moderate and severe oral mucositis.
* Subject is able (in the investigator's opinion) and willing to comply with all study requirements.
* Subject is willing and able to communicate with the investigator.
* Subject has acceptable haematological and biochemical function, in the opinion of the investigator, as demonstrated by appropriate laboratory parameter levels including liver and renal function (estimated glomerular filtration rate as measured by the Cockcroft-Gault formula >0.5 lower limit of normal, aspartate aminotransferase/alanine aminotransferase <2.5 the upper limit of normal (ULN) and bilirubin <1.5 ULN), and in the opinion of the investigator, acceptable bone marrow reserve.
* Vital signs at screening (after five minutes resting measured in the supine position) must be within the following ranges:

  i. Body temperature between 35.0-37.5°C ii. Systolic blood pressure, 90-150 mmHg iii. Diastolic blood pressure, 60-90 mmHg iv. Pulse rate, 40-99 beats per minute Blood pressure and pulse rate will be taken again in a standing position. After two minutes standing, there shall be no more than a 20 mmHg drop in systolic or 10 mmHg drop in diastolic blood pressure, associated with clinical manifestation of postural hypotension.
* Subject has an Eastern Co-operative Oncology Group Performance Status of 0, 1 or 2.
* Subject is willing for his or her name to be notified to the responsible authorities for participation in this study, as applicable in individual countries.
* Subject is willing to allow his or her primary care practitioner and consultant to be notified of participation in the study.

Exclusion Criteria:

* Subjects undergoing chemotherapy only.
* Subjects with cancer other than HNSCC as the primary tumour.
* Subjects who have undergone reconstructive oral surgery for HNSCC (within the last eight weeks).
* Subjects with RTOG Grade 4 oral mucositis (necrosis or deep ulceration, with or without bleeding).
* Subjects requiring hospital admission or extended hospitalisation for total parenteral nutrition, intravenous analgesia and/or intravenous antibiotics for the treatment of oral mucositis.
* Subjects with aphthous stomatitis, herpetic mucositis, oral thrush, denture/oral trauma, gangrenous stomatitis, acute necrotising stomatitis or other oral condition that may in the opinion of the investigator affect the oromucosal absorption of Sativex® in the absence of oral mucositis.
* Any surgical or medical condition, significant disease or disorder or any finding on physical examination (or oral examination) (other than their underlying condition) which might significantly alter the absorption, distribution, metabolism or excretion of drugs or that, in the opinion of the investigator, may put the subject at risk, influence the result of the study, or the subjects' ability to participate in the study.
* Clinical evidence of acute or chronic liver disease or liver injury as indicated by clinically significant abnormal liver function tests such as aspartate aminotransferase, alanine aminotransferase, gamma glutamyl-transpeptidase, alkaline phosphatase, (any ≥2.5 ULN ) or serum bilirubin (≥1.5 ULN) unless there is another more likely explanation (e.g. Gilbert's syndrome).
* Any change in medication within 14 days prior to dosing and throughout the study which might significantly alter the absorption, distribution, metabolism or excretion of the investigational medicinal product (IMP), in the opinion of the investigator.
* History of drug abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.
* Any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP(s).
* Positive result for the presence of hepatitis B surface antigen, hepatitis C virus antibodies, or human immunodeficiency virus antibodies.
* Currently using or has used cannabis, cannabinoid-based medications (e.g. Marinol®, Nabilone®, Cannador®) or Acomplia® (rimonabant) or taranabant within 30 days of study entry and unwilling to abstain for the duration of the study.
* Any known or suspected history or family history of schizophrenia, or other psychotic illness, history of severe personality disorder or other severe significant psychiatric disorder other than depression associated with underlying condition.
* Any history of epilepsy as evidenced by one or more seizures in the last 12 months.
* Significant cardiac disease, or has a cardiac disorder that in the opinion of the investigator would put the subject at risk of a clinically relevant arrhythmia or myocardial infarction, or has a secondary or tertiary atrioventricular block, or evidence of clinically significant cardiac disease on electrocardiogram at screening.
* Female subjects of child bearing potential and male subjects whose partner is of child bearing potential, unless willing to ensure that they or their partner use two effective forms of contraception, for example, oral contraception, double barrier, intra-uterine device, during the study and for three months thereafter (Note: a male condom should not be used in conjunction with a female condom).
* Female subjects who are pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter.
* Subjects who have received an IMP within the 12 weeks prior to the screening visit.
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the result of the study, or the subject's ability to participate in the study.
* Following a physical examination, the subject has any abnormalities that, in the opinion of the investigator would prevent the subject from safe participation in the study.
* Unwilling to abstain from donation of blood during the study.
* Travel outside the country of residence planned during the study.
* Subjects previously enrolled into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The time to peak plasma concentration (Cmax) of THC, 11-hydroxy-THC, CBD, 7-hydroxy-CBD and 6-hydroxy-CBD after a single dose of Sativex | Pre-dose then 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours post-dose
  Blood samples for PK analysis were taken at pre-defined time-points by either direct venipuncture or an indwelling cannula inserted in a forearm vein. Blood was drawn from each subject into a five-mL lithium-heparinised tube. The allowable window for sample collection was ±5 minutes at all PK time points with the exception of 8 hours (window of ±1 hour) and 24 hours (±2 hours).
Area under the concentration-time curve from administration until the last sampling point (t) equal or above the Lower Limit of Quantification (AUC(0-t)) of THC, 11-hydroxy-THC, CBD, 7-hydroxy-CBD and 6-hydroxy-CBD after a single dose of Sativex | Pre-dose then 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours post-dose
  Blood samples for PK analysis were taken at pre-defined time-points by either direct venipuncture or an indwelling cannula inserted in a forearm vein. Blood was drawn from each subject into a five-mL lithium-heparinised tube. The allowable window for sample collection was ±5 minutes at all PK time points with the exception of 8 hours (window of ±1 hour) and 24 hours (±2 hours).
Area under the concentration-time curve extrapolated to infinity (AUC(0-∞)) of THC, 11-hydroxy-THC, CBD, 7-hydroxy-CBD and 6-hydroxy-CBD after a single dose of Sativex | Pre-dose then 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours post-dose
  Blood samples for PK analysis were taken at pre-defined time-points by either direct venipuncture or an indwelling cannula inserted in a forearm vein. Blood was drawn from each subject into a five-mL lithium-heparinised tube. The allowable window for sample collection was ±5 minutes at all PK time points with the exception of 8 hours (window of ±1 hour) and 24 hours (±2 hours).

SECONDARY OUTCOMES:
Median time to maximum plasma concentration (Tmax) of THC, 11-hydroxy-THC, CBD, 7-hydroxy-CBD and 6-hydroxy-CBD after a single dose of Sativex | Pre-dose then 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours post-dose
  Blood samples for PK analysis were taken at pre-defined time-points by either direct venipuncture or an indwelling cannula inserted in a forearm vein. Blood was drawn from each subject into a five-mL lithium-heparinised tube. The allowable window for sample collection was ±5 minutes at all PK time points with the exception of 8 hours (window of ±1 hour) and 24 hours (±2 hours).
Terminal half-life (t1/2) of THC, 11-hydroxy-THC, CBD, 7-hydroxy-CBD and 6-hydroxy-CBD after a single dose of Sativex | Pre-dose then 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours post-dose
  Blood samples for PK analysis were taken at pre-defined time-points by either direct venipuncture or an indwelling cannula inserted in a forearm vein. Blood was drawn from each subject into a five-mL lithium-heparinised tube. The allowable window for sample collection was ±5 minutes at all PK time points with the exception of 8 hours (window of ±1 hour) and 24 hours (±2 hours).
Apparent total body clearance of drug from plasma (CL/F) of THC, 11-hydroxy-THC, CBD, 7-hydroxy-CBD and 6-hydroxy-CBD after a single dose of Sativex | Pre-dose then 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours post-dose
  Blood samples for PK analysis were taken at pre-defined time-points by either direct venipuncture or an indwelling cannula inserted in a forearm vein. Blood was drawn from each subject into a five-mL lithium-heparinised tube. The allowable window for sample collection was ±5 minutes at all PK time points with the exception of 8 hours (window of ±1 hour) and 24 hours (±2 hours).
The incidence of adverse events as a measure of subject safety | Day 1 - Day 30
  The numbers of subjects who experienced an adverse event during the study is presented.

CONTACTS AND LOCATIONS:
Overall Officials: James Ritter, DPhil FRCP FMedSci, Study Chair — Quintiles Drug Research Unit at Guy's Hospital
Locations (1):
- Quintiles London Drug Research Unit, London, United Kingdom